CLINICAL TRIAL: NCT05420194
Title: Assessment of Postural Stability in Patients With Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Collaborators: Marmara University (Other)
Responsible Party: Principal Investigator, Özgül Öztürk, Assistant Professor, Acibadem University
Other Study IDs: ATADEK -2022/7
Record Dates: First submitted 2022-06-12; First posted 2022-06-15 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Knee Arthritis; Arthroplasty Complications; Obesity; Balance; Distorted
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Postural stability measurement — Postural stability of the participants will be evaluated with the NeuroCom Balance Master Static Posturography device. Evaluations will be carried out in the presence of two physiotherapists to prevent the patient from falling. Posturography devices allow us to quantitatively evaluate posture and balance and obtain objective results by measuring postural sway.
Other: Timed Up and Go test — During the Timed Up and Go test, which is applied to evaluate dynamic balance and performance, the participant is asked to get up from the chair, walk 3 meters and sit back on the chair. The participant's time to complete the test is recorded. Completion of the test for more than 10 seconds indicates an increased risk of falling

SUMMARY:
Postural balance can be described as the integration of the information obtained from visual, vestibular and somatosensory systems. Postural stability is achieved by sensory information about the static or dynamic position of the body resulting in an appropriate motor response. Poor postural stability in individuals with knee osteoarthritis often results in an increased risk of falling and decrease in mobility. It has been reported that 40% of knee osteoarthritis patients fall at least once in a year. Total knee arthroplasty (TKA) is a surgical treatment approach applied to individuals with advanced knee osteoarthritis. It has been shown that this method provides an improvement in the postural stability levels of individuals compared to the preoperative period and a decrease in number of falls reported by the patient. Even if this improvement is achieved, postural stability losses can still be observed in individuals undergoing TKA which affect balance performance.

Obesity is defined by an excessive increase in the ratio of body fat mass relative to lean mass. Individuals with a Body Mass Index (BMI) above 30 kg/m2 are defined as obese. Changes in body composition and increased adiposity rate lead to significant locomotor system problems. A decrease in postural control, increased risk of falling or fear of falling can be defined as locomotor system problems. It has been reported that there is a relationship between increased fat ratio and loss of postural stability in adult obese individuals.

In a published study, it was reported that as of 2029, 46% of the population in America will be obese or morbidly obese, and 69% of individuals who have undergone total knee arthroplasty surgery will be obese or morbidly obese. Obesity causes several complications such as increased mortality and increase in likelihood of revision surgery that can be seen after total knee arthroplasty. Therefore, it is clinically important to determine the functional status and balance status in order to reduce the possible long-term complications that may develop in the post-operative period and the risk of falling, especially in obese individuals.

The effects of increasing obesity level on postural stability in individuals undergoing total knee arthroplasty are unknown. In this context, the aim of our study is to compare the postural stability levels of normal, overweight and obese individuals who underwent total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Follow-up period is between 1-5 years,
* Volunteer to participate in the study,

Exclusion Criteria:

* Having undergone revision surgery on the same or opposite knee after total knee arthroplasty,

  - Presence of vertigo or another neurological disease,
* Patients who have undergone total hip replacement.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had undergone total knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Postural Stability | Day 1
  Postural stability of the participants will be evaluated with the NeuroCom Balance Master Static Posturography device. Posturography devices allow us to quantitatively evaluate posture and balance and obtain objective results by measuring postural sway. Sensory impairment, motor impairment and functional limitations can be evaluated with this device. In the study, the Clinical Test of Sensory Interaction on Balance (mCTSIB) will be used to evaluate the sensory status, and the Limits of Stability-LOS Test, Rhythmic Weight Shift-RWS will be used to evaluate the motor status. The Unilateral Stance-US Test will also be used to evaluate the functional limitation.
Falls Efficacy Scale | Day 1
  Falls Efficacy Scale measures fear of falling during different social or physical activities at home and outside with a scale consisting of 16 questions. The total score ranges from 16 to 64, and a high score indicates greater fear of falling.

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Day 1
  SPPB was developed to measure the strength and performance of the lower extremity muscles. Walking speed, standing balance and getting up from a chair for 5 times are the sub-components of this test. For standing balance, the patient will be asked to hold his position for 10 seconds in normal, semi-tandem and tandem foot postures. For walking speed, walking time of 4 m distance will be recorded. Finally, the time the participant sit to stand for 5 times from a chair without arm support will be recorded.
Timed Up and Go Test | Day 1
  The Timed Up and Go test is applied to evaluate dynamic balance and performance. During this test the participant will be asked to get up from the chair, walk 3 meters and sit back on the chair. The participant's time to complete the test is recorded. Completion of the test for more than 10 seconds indicates an increased risk of falling.
Pain Severity | Day 1
  The pain intensity felt by the participants at rest and during movement will be evaluated with the Visual Analog Scale. Visual Analog Scale determines pain severity with a 10 cm horizontal line and "0" indicates no pain, "10" indicates unbearable pain. The point marked by the patient on this line will be measured and recorded with the help of a ruler.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Acıbadem University, Istanbul
  - Marmara University, Istanbul